CLINICAL TRIAL: NCT01730040
Title: A Randomized, Double-Blind Study of the Efficacy and Safety of Alirocumab Added on to Atorvastatin Versus Ezetimibe Added on to Atorvastatin Versus Atorvastatin Dose Increase Versus Switch to Rosuvastatin in Patients Who Are Not Controlled on Atorvastatin
Brief Title: Study of the Efficacy and Safety of Alirocumab (REGN727/SAR236553) in Combination With Other Lipid-modifying Treatment (LMT) (ODYSSEY OPTIONS I)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R727-CL-1110
Record Dates: First submitted 2012-11-09; First posted 2012-11-21 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-07

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Atorvastatin; Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Atorvastatin 40 mg (Active Comparator): Participants, who were receiving atorvastatin 20 mg over-encapsulated tablets orally at baseline, received atorvastatin 40 mg over-encapsulated tablets orally once daily (QD), placebo for alirocumab SC injection every two weeks (Q2W), and placebo for ezetimibe over-encapsulated tablets orally QD added to stable Lipid-Modifying Therapy (LMT) for 24 weeks.
  Interventions: Drug: Atorvastatin; Drug: Placebo
- Ezetimibe 10 mg + Atorvastatin 20 mg (Active Comparator): Participants, who were receiving atorvastatin 20 mg over-encapsulated tablets orally at baseline, received ezetimibe 10 mg over-encapsulated tablets orally QD, atorvastatin 20 mg over-encapsulated tablets orally QD, and placebo for alirocumab SC injection Q2W added to stable LMT for 24 weeks.
  Interventions: Drug: Atorvastatin; Drug: Ezetimibe; Drug: Placebo
- Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg (Experimental): Participants, who were receiving atorvastatin 20 mg over-encapsulated tablets orally at baseline, received Alirocumab 75 mg SC injection Q2W, atorvastatin 20 mg over-encapsulated tablets orally QD, and placebo for ezetimibe over-encapsulated tablets orally QD added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on baseline disease characteristic and medical history.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin; Drug: Placebo
- Atorvastatin 80 mg (Active Comparator): Participants, who were receiving atorvastatin 40 mg over-encapsulated tablets orally at baseline, received Atorvastatin 80 mg over-encapsulated tablets orally QD, placebo for alirocumab SC injection Q2W, and placebo for ezetimibe over-encapsulated tablets orally QD added to stable LMT for 24 weeks.
  Interventions: Drug: Atorvastatin; Drug: Placebo
- Rosuvastatin 40 mg (Active Comparator): Participants, who were receiving atorvastatin 40 mg over-encapsulated tablets orally at baseline, received rosuvastatin 40 mg over-encapsulated tablets orally QD, placebo for alirocumab SC injection Q2W, and placebo for ezetimibe over-encapsulated tablets orally QD added to stable LMT for 24 weeks.
  Interventions: Drug: Rosuvastatin; Drug: Placebo
- Ezetimibe 10 mg + Atorvastatin 40 mg (Active Comparator): Participants, who were receiving atorvastatin 40 mg over-encapsulated tablets orally at baseline, received ezetimibe 10 mg over-encapsulated tablets orally QD, atorvastatin 40 mg over-encapsulated tablets orally QD, and placebo for alirocumab SC injection Q2W added to stable LMT for 24 weeks.
  Interventions: Drug: Atorvastatin; Drug: Ezetimibe; Drug: Placebo
- Alirocumab 75 mg/ up to 150 mg + Atorvastatin 40 mg (Experimental): Participants, who were receiving atorvastatin 40 mg over-encapsulated tablets orally at baseline, received alirocumab 75 mg SC injection Q2W, atorvastatin 40 mg over-encapsulated tablets orally QD, and placebo for ezetimibe over-encapsulated tablets orally QD added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on baseline disease characteristic and medical history.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Alirocumab — Alirocumab administered as a SC injection of 1 mL into the abdomen, thigh, or outer area of the upper arm.
  Other Names: REGN727/SAR236553
  Arms: Alirocumab 75 mg/ up to 150 mg + Atorvastatin 40 mg; Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg
Drug: Atorvastatin — Atorvastatin over-encapsulated tablets orally.
  Arms: Alirocumab 75 mg/ up to 150 mg + Atorvastatin 40 mg; Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Atorvastatin 40 mg; Atorvastatin 80 mg; Ezetimibe 10 mg + Atorvastatin 20 mg; Ezetimibe 10 mg + Atorvastatin 40 mg
Drug: Ezetimibe — Ezetimibe over-encapsulated tablet orally.
  Other Names: Ezetrol
  Arms: Ezetimibe 10 mg + Atorvastatin 20 mg; Ezetimibe 10 mg + Atorvastatin 40 mg
Drug: Rosuvastatin — Rosuvastatin over-encapsulated tablets orally.
  Other Names: Crestor
  Arms: Rosuvastatin 40 mg
Drug: Placebo — Placebo for alirocumab and ezetimibe.

SUMMARY:
This is a randomized, double-blind, active-comparator, parallel-group study in patients at high cardiovascular risk with nonfamilial hypercholesterolemia or heterozygous familial hypercholesterolemia (heFH).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with screening (visit 1) LDL-C greater than or equal to 70 mg/dL with documented CVD, not adequately controlled with a daily dose of atorvastatin. OR
2. Patients with screening (visit 1) LDL-C greater than or equal to 100 mg/dL at high risk for CVD who are not adequately controlled with a daily dose of atorvastatin.

Exclusion Criteria:

1. LDL-C greater than 250 mg/dL
2. LDL-C less than 70 mg/dL at the screening visit in patients with history of documented CVD
3. LDL-C less than 100 mg/dL at the screening visit in patients without history of documented CHD or non-CHD CVD, but with other risk factors
4. TG greater than 400 mg/dL
5. Homozygous FH (clinically or previous genotyping)
6. Currently taking a statin that is not atorvastatin
7. Currently taking Ezetimibe (EZE)
8. Not on a stable dose of allowable lipid modifying treatments (LMT)

(The inclusion/ exclusion criteria provided above is not intended to contain all considerations relevant to a patient's potential participation in this clinical trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (97):
- United States (56):
  - Mobile, Alabama
  - Chandler, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Beverly Hills, California
  - Lakeland Village, California
  - Newport Beach, California
  - Northridge, California
  - Sacramento, California
  - Walnut Creek, California
  - Milford, Connecticut
  - Atlantis, Florida
  - Boca Raton, Florida
  - Clearwater, Florida
  - Jacksonville, Florida
  - Miami (2 Locations), Florida
  - Oviedo, Florida
  - Pinellas Park, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Boise, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Morton, Illinois
  - Indianapolis, Indiana
  - Newton, Kansas
  - Overland Park, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Auburn, Maine
  - Bethesda, Maryland
  - Edina, Minnesota
  - Rochester, Minnesota
  - Olive Branch, Mississippi
  - Port Gibson, Mississippi
  - St Louis, Missouri
  - Butte, Montana
  - Las Vegas, Nevada
  - Williamsville, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Warwick, Rhode Island
  - Greer, South Carolina
  - Summerville, South Carolina
  - Kingsport, Tennessee
  - Dallas (2 Locations), Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Bountiful, Utah
  - Marion, Utah
  - Salt Lake City, Utah
  - Renton, Washington
- Australia (5):
  - Herston QLD
  - New Lambton Heights
  - Perth
  - Sherwood
  - Woolloongabba
- Canada (7):
  - Brampton, Ontario
  - Etobicoke, Ontario
  - London, Ontario
  - Newmarke, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
- France (3):
  - Dijon
  - Lille
  - Vénissieux
- Germany (6):
  - Bad Oeynhausen
  - Berlin
  - Cologne
  - Munich
  - Regensburg
  - Ulm
- Italy (5):
  - Chiete
  - Genova
  - Napoli
  - Palermo
  - Roma (2 Locations)
- Mexico (6):
  - Distrito Federal
  - Guadalajara
  - Guadalajara, Jalisco
  - Monterrey Nuevo Leon
  - Tijuana Baja California
  - Zapopan Jalisco
- Spain (3):
  - Barcelona (3 Locations)
  - Madrid
  - Sant Joan Despí
- United Kingdom (6):
  - Carmarthen
  - Chester
  - Peterborough
  - Salford
  - Stevenage
  - West Bromwich, West Midlands

REFERENCES:
- [Derived] Mahmood T, Minnier J, Ito MK, Li QH, Koren A, Kam IW, Fazio S, Shapiro MD. Discordant responses of plasma low-density lipoprotein cholesterol and lipoprotein(a) to alirocumab: A pooled analysis from 10 ODYSSEY Phase 3 studies. Eur J Prev Cardiol. 2021 Jul 23;28(8):816-822. doi: 10.1177/2047487320915803. Epub 2020 Apr 10. PMID 34298554
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Ray KK, Ginsberg HN, Davidson MH, Pordy R, Bessac L, Minini P, Eckel RH, Cannon CP. Reductions in Atherogenic Lipids and Major Cardiovascular Events: A Pooled Analysis of 10 ODYSSEY Trials Comparing Alirocumab With Control. Circulation. 2016 Dec 13;134(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.116.024604. Epub 2016 Oct 24. PMID 27777279
- [Derived] Bays H, Gaudet D, Weiss R, Ruiz JL, Watts GF, Gouni-Berthold I, Robinson J, Zhao J, Hanotin C, Donahue S. Alirocumab as Add-On to Atorvastatin Versus Other Lipid Treatment Strategies: ODYSSEY OPTIONS I Randomized Trial. J Clin Endocrinol Metab. 2015 Aug;100(8):3140-8. doi: 10.1210/jc.2015-1520. Epub 2015 Jun 1. PMID 26030325
- [Derived] Robinson JG, Colhoun HM, Bays HE, Jones PH, Du Y, Hanotin C, Donahue S. Efficacy and safety of alirocumab as add-on therapy in high-cardiovascular-risk patients with hypercholesterolemia not adequately controlled with atorvastatin (20 or 40 mg) or rosuvastatin (10 or 20 mg): design and rationale of the ODYSSEY OPTIONS Studies. Clin Cardiol. 2014 Oct;37(10):597-604. doi: 10.1002/clc.22327. Epub 2014 Sep 30. PMID 25269777

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 85 sites in 9 countries. Overall, 859 subjects were screened between 24 October 2012 and 26 September 2013, 504 of whom were screen failures. Screen failures ware mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to prior history of myocardial infarction or ischemic stroke, and intensity of statin treatment (atorvastatin 20 or 40 mg). Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:1:1:1:1:1:1 ratio after confirmation of selection criteria.
Groups:
- Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg: Participants, who were receiving atorvastatin 40 mg over-encapsulated tablets orally at baseline, received alirocumab 75 mg SC injection Q2W, atorvastatin 40 mg over-encapsulated tablets orally QD, and placebo for ezetimibe over-encapsulated tablets orally QD added to stable LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on baseline disease characteristic and medical history.
Period: Overall Study
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Started | 57 | 55 | 57 | 47 | 45 | 47 | 47
Treated | 57 | 55 | 57 | 47 | 45 | 46 | 47
Completed | 44 | 40 | 46 | 39 | 39 | 40 | 38
Not Completed | 13 | 15 | 11 | 8 | 6 | 7 | 9
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Subject moved | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Other than specified | 7 | 8 | 5 | 5 | 5 | 4 | 4
Not completed — Adverse Event | 4 | 3 | 5 | 3 | 1 | 1 | 2
Not completed — Poor compliance to protocol | 2 | 4 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/ up to 150 mg + Atorvastatin 40 mg | Total
Number analyzed (Participants) | 57 | 55 | 57 | 47 | 45 | 47 | 47 | 355
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.91) | 65.7 (8.96) | 62.2 (10.03) | 63.2 (10.89) | 57.5 (9.96) | 63.9 (10.33) | 64.2 (10.36) | 62.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 24 | 14 | 13 | 11 | 16 | 124
  Male | 35 | 31 | 33 | 33 | 32 | 36 | 31 | 231
Low density lipoprotein cholesterol (LDL-C) in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C from Friedewald formula.
  mg/dL | 100.3 (29.8) | 100.4 (29.5) | 103.9 (34.9) | 108.6 (37.5) | 109.8 (39.0) | 98.9 (29.2) | 116.4 (37.4) | 105.1 (34.1)
LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] — Calculated LDL-C from Friedewald formula.
  mmol/L | 2.957 (0.773) | 2.599 (0.765) | 2.692 (0.905) | 2.813 (0.97) | 2.844 (1.011) | 2.562 (0.756) | 3.016 (0.968) | 2.723 (0.884)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-treat (ITT) Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -5 (4.6) | -20.5 (4.7) | -44.1 (4.5) | -4.8 (4.2) | -21.4 (4.2) | -22.6 (4.3) | -54 (4.3)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Alirocumab group was compared to the corresponding active control group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Threshold for significance ≤ 0.01; LS Mean Difference = -39.1, 99% CI 2-sided [-55.9 to -22.2]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; As described in statistical analysis 1 of the endpoint; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -23.6, 99% CI 2-sided [-40.7 to -6.5]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -49.2, 99% CI 2-sided [-65 to -33.5]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -32.6, 99% CI 2-sided [-48.4 to -16.9]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -31.4, 99% CI 2-sided [-47.4 to -15.4]

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule [whatever atorvastatin, rosuvastatin or ezetimibe], whichever came first) (on-treatment analysis).
Time Frame: From Baseline to Week 24
Population: Modified ITT (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 52 | 52 | 52 | 47 | 45 | 46 | 46
percent change | -6.1 (4.6) | -23.7 (4.7) | -48.6 (4.5) | -5.0 (4.4) | -22.9 (4.4) | -24.5 (4.5) | -57.8 (4.5)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 1% level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -42.5, 99% CI 2-sided [-59.2 to -25.7]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — Threshold for significance≤ 0.01; LS Mean Difference = -24.9, 99% CI 2-sided [-41.9 to -7.8]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -52.8, 99% CI 2-sided [-69.2 to -36.5]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Threshold for significance ≤ 0.01; LS Mean Difference = -35.0, 99% CI 2-sided [-51.3 to -18.6]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -33.4, 99% CI 2-sided [-50.0 to -16.8]

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -8.5 (3.9) | -22.6 (3.9) | -48.4 (3.8) | -14.5 (3.2) | -23.3 (3.2) | -29.7 (3.2) | -50.5 (3.2)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -39.8, 99% CI 2-sided [-54 to -25.6]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -25.8, 99% CI 2-sided [-40.0 to -11.6]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -36.0, 99% CI 2-sided [-47.7 to -24.3]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -27.3, 99% CI 2-sided [-39.2 to -15.4]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -20.9, 99% CI 2-sided [-32.8 to -8.9]

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-Treatment Analysis
Description: Calculated LDL-C values were obtained from Friedewald formula. Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule [whatever atorvastatin, rosuvastatin or ezetimibe], whichever came first) (on-treatment analysis).
Time Frame: From Baseline to Week 24
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 52 | 52 | 52 | 47 | 45 | 46 | 46
percent change | -9.2 (3.1) | -27.1 (3.1) | -53.7 (3.1) | -14.6 (3.2) | -23.3 (3.2) | -30.7 (3.2) | -50.9 (3.2)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -44.5, 99% CI 2-sided [-55.8 to -33.1]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -26.6, 99% CI 2-sided [-38.0 to -15.2]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -36.3, 99% CI 2-sided [-48.1 to -24.5]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -27.7, 99% CI 2-sided [-39.6 to -15.8]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -20.2, 99% CI 2-sided [-32.2 to -8.2]

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 51 | 50 | 53 | 45 | 44 | 45 | 42
percent change | -4.4 (3.5) | -10.1 (3.6) | -33.7 (3.4) | -3.5 (3.3) | -10.9 (3.2) | -14.3 (3.3) | -41.9 (3.4)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -29.3, 99% CI 2-sided [-42.0 to -16.6]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -23.6, 99% CI 2-sided [-36.6 to -10.7]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -38.4, 99% CI 2-sided [-50.8 to -26.0]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -30.9, 99% CI 2-sided [-43.2 to -18.6]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -27.6, 99% CI 2-sided [-40.1 to -15.1]

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (ie. up to 21 days after last injection or 3 days after the last capsule [whatever atorvastatin, rosuvastatin or ezetimibe], whichever came first).
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the mITT population with one baseline and at least one post-baseline Apo B value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 48 | 47 | 50 | 44 | 44 | 44 | 41
percent change | -5.1 (3.3) | -12.6 (3.5) | -37.7 (3.2) | -4.4 (3.4) | -12.8 (3.4) | -16.3 (3.4) | -42.7 (3.5)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -32.6, 99% CI 2-sided [-44.6 to -20.6]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -25.1, 99% CI 2-sided [-37.3 to -12.8]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -38.3, 99% CI 2-sided [-51.2 to -25.4]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -29.8, 99% CI 2-sided [-42.6 to -17.1]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -26.4, 99% CI 2-sided [-39.4 to -13.4]

7. Secondary Outcome: Percent Change From Baseline in Non-High-density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -6.3 (3.9) | -15.1 (4.0) | -36.7 (3.9) | -6.5 (3.6) | -17.4 (3.6) | -21.0 (3.7) | -47.6 (3.7)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -30.4, 99% CI 2-sided [-44.7 to -16.1]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -21.6, 99% CI 2-sided [-36.1 to -7.1]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -41.1, 99% CI 2-sided [-54.7 to -27.5]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -30.2, 99% CI 2-sided [-43.7 to -16.6]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -26.6, 99% CI 2-sided [-40.3 to -12.8]

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection or 3 days after the last capsule [whatever atorvastatin, rosuvastatin or ezetimibe], whichever came first).
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the mITT population with one baseline and at least one post-baseline Non-HDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 52 | 52 | 52 | 47 | 45 | 46 | 46
percent change | -7.5 (3.8) | -18.1 (4.0) | -40.5 (3.7) | -7.0 (3.7) | -18.4 (3.7) | -23.3 (3.8) | -50.5 (3.8)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -33.0, 99% CI 2-sided [-47.0 to -19.0]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -22.4, 99% CI 2-sided [-36.6 to -8.1]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -43.6, 99% CI 2-sided [-57.4 to -29.7]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -32.1, 99% CI 2-sided [-46.0 to -18.3]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -27.3, 99% CI 2-sided [-41.4 to -13.2]

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline Total-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -4.0 (2.7) | -11.2 (2.8) | -27.1 (2.7) | -4.8 (2.8) | -11.7 (2.8) | -15.2 (2.9) | -33.6 (2.9)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -23.1, 99% CI 2-sided [-32.9 to -13.2]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -15.8, 99% CI 2-sided [-25.8 to -5.8]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -28.9, 99% CI 2-sided [-39.4 to -18.4]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -21.9, 99% CI 2-sided [-32.4 to -11.4]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -18.4, 99% CI 2-sided [-29.1 to -7.7]

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 51 | 50 | 53 | 45 | 44 | 45 | 42
percent change | -6.9 (2.8) | -13.1 (2.8) | -38.4 (2.7) | -9.5 (2.5) | -14.1 (2.5) | -20.3 (2.5) | -36.2 (2.5)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -31.5, 99% CI 2-sided [-41.6 to -21.3]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -25.3, 99% CI 2-sided [-35.4 to -15.2]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -26.7, 99% CI 2-sided [-35.9 to -17.5]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -22.2, 99% CI 2-sided [-31.5 to -12.9]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -15.9, 99% CI 2-sided [-25.2 to -6.6]

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 24
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -7.1 (3.2) | -17.2 (3.2) | -40.6 (3.2) | -13.0 (2.6) | -19.8 (2.7) | -27.5 (2.7) | -42.3 (2.7)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -33.5, 99% CI 2-sided [-45.3 to -21.6]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -23.4, 99% CI 2-sided [-35.2 to -11.6]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -29.3, 99% CI 2-sided [-39.0 to -19.6]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -22.5, 99% CI 2-sided [-32.3 to -12.7]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -14.8, 99% CI 2-sided [-24.7 to -4.9]

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 24
Population: Total-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -6.5 (2.4) | -13.2 (2.4) | -29.0 (2.4) | -9.9 (2.1) | -13.5 (2.1) | -19.2 (2.1) | -29.0 (2.1)
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -22.6, 99% CI 2-sided [-31.4 to -13.8]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -15.8, 99% CI 2-sided [-24.6 to -7.0]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -19.1, 99% CI 2-sided [-26.9 to -11.4]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -15.4, 99% CI 2-sided [-23.3 to -7.6]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = -9.8, 99% CI 2-sided [-17.7 to -1.9]

13. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 were obtained from a multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to week 24 regardless of status on- or off-treatment were included in the imputation model (ITT analysis).
Time Frame: Up to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percentage of participants | 34.5 | 68.4 | 87.2 | 18.5 | 62.2 | 65.1 | 84.6
Statistical Analysis 1: Comparison: Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant). Statistical analysis used a multiple imputation approach followed by a Logistic regression model; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 16.7, 99% CI 2-sided [3.9 to 71.7]
Statistical Analysis 2: Comparison: Ezetimibe 10 mg + Atorvastatin 20 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0284, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 3.4, 99% CI 2-sided [0.8 to 14.6]
Statistical Analysis 3: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 83.2, 99% CI 2-sided [11.6 to 596.8]
Statistical Analysis 4: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0025, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 7.2, 99% CI 2-sided [1.3 to 38.3]
Statistical Analysis 5: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0011, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 9.1, 99% CI 2-sided [1.6 to 52.2]

14. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 were obtained from a multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 24 i.e. up to 21 days after last injection or 3 days after the last capsule [whatever atorvastatin, rosuvastatin or ezetimibe], whichever came first (on-treatment analysis).
Time Frame: Up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 52 | 52 | 52 | 47 | 45 | 46 | 46
percentage of participants | 37.8 | 72.2 | 91.2 | 18.5 | 64.0 | 66.2 | 90.0
Statistical Analysis 1: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant) for atorvastatin 40 mg baseline stratification). Statistical analysis used a multiple imputation approach followed by a Logistic regression model; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 128.4, 99% CI 2-sided [14.2 to 1157]
Statistical Analysis 2: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0015, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 10.9, 99% CI 2-sided [1.6 to 75.4]
Statistical Analysis 3: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0008, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 13.7, 99% CI 2-sided [1.8 to 101.1]

15. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: as for outcome 13
Time Frame: Up to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percentage of participants | 16.0 | 50.3 | 79.2 | 10.2 | 42.2 | 54.2 | 77.2
Statistical Analysis 1: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 116.8, 99% CI 2-sided [14.7 to 927.5]
Statistical Analysis 2: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 13.2, 99% CI 2-sided [2.5 to 68.8]
Statistical Analysis 3: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0004, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 9.9, 99% CI 2-sided [1.9 to 51.9]

16. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-Treatment Analysis
Description: as for outcome 14
Time Frame: Up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 52 | 52 | 52 | 47 | 45 | 46 | 46
percentage of participants | 20.0 | 55.1 | 82.3 | 10.5 | 42.4 | 55.3 | 83.7
Statistical Analysis 1: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 162.1, 99% CI 2-sided [17.3 to 1520.5]
Statistical Analysis 2: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 19.8, 99% CI 2-sided [3.1 to 126.3]
Statistical Analysis 3: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p = 0.0002, Regression, Logistic — Threshold for significance ≤ 0.01; Odds Ratio (OR) = 13.9, 99% CI 2-sided [2.2 to 88.1]

17. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from from a multiple imputation approach model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -20.2 (4.0) | -10.6 (4.4) | -23.6 (4.0) | -9.7 (4.1) | -4.9 (3.7) | 0.2 (3.9) | -30.8 (4.1)
Statistical Analysis 1: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant) for atorvastatin 40 mg baseline stratification). Statistical analysis used a multiple imputation approach followed by a robust regression model; Test type: Superiority or Other; p = 0.0004, Regression, Robust — Threshold for significance ≤ 0.01; Adjusted Mean Difference = -21.1, 99% CI 2-sided [-36.3 to -5.9]
Statistical Analysis 2: Comparison: Rosuvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.01; Adjusted Mean Difference = -25.9, 99% CI 2-sided [-40.2 to -11.6]
Statistical Analysis 3: Comparison: Ezetimibe 10 mg + Atorvastatin 40 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Analysis description as per the statistical analysis 1 of this endpoint; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.01; Adjusted Mean Difference = -31.0, 99% CI 2-sided [-45.6 to -16.4]

18. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | 1.9 (2.0) | -0.1 (2.1) | 4.8 (2.0) | 4.7 (2.7) | 5.7 (2.7) | 2.0 (2.7) | 7.7 (2.7)
Statistical Analysis 1: Comparison: Atorvastatin 80 mg vs Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant) for atorvastatin 40 mg baseline stratification); Test type: Superiority or Other; p = 0.4456, Mixed Models Analysis — Threshold for significance ≤ 0.01; LS Mean Difference = 2.9, 99% CI 2-sided [-7.0 to 12.9]

19. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: as for outcome 17
Time Frame: From Baseline to Week 24
Population: ITT population: all randomized and treated participants with one baseline and at least one post-baseline fasting triglycerides value on- or off-treatment.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -6.7 (3.7) | -3.3 (4.1) | -12.0 (3.7) | -7.3 (4.1) | -0.5 (4.0) | -13.9 (4.1) | -19.1 (4.10)

20. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 51 | 50 | 53 | 45 | 44 | 45 | 42
percent change | 1.2 (1.5) | 1.0 (1.6) | 7.6 (1.5) | 2.2 (2.0) | 4.7 (1.9) | -1.8 (1.9) | 5.8 (2.0)

21. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from from a multiple imputation approach model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Lipoprotein (a) ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -11.7 (4.0) | -5.4 (4.0) | -24.0 (4.0) | -1.6 (4.5) | 11.5 (4.6) | 7.9 (4.5) | -27.9 (4.5)

22. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 24
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -3.2 (1.8) | -1.7 (1.8) | 4.1 (1.8) | 3.0 (2.6) | 4.6 (2.7) | 4.6 (2.7) | 8.5 (2.7)

23. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: as for outcome 21
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 53 | 53 | 55 | 47 | 45 | 46 | 46
percent change | -4.7 (4.2) | 0.5 (4.2) | -12.4 (4.2) | -4.6 (4.0) | -3.7 (4.1) | -16.8 (4.0) | -12.1 (4.0)

24. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 24
Population: Apo A-1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Number analyzed (Participants) | 51 | 50 | 53 | 45 | 44 | 45 | 42
percent change | -0.8 (1.5) | 1.7 (1.4) | 5.4 (1.4) | 1.6 (1.7) | 5.6 (1.7) | 1.6 (1.7) | 9.4 (1.7)

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 24
Description: Treatment emergent adverse events that developed during on¬-treatment period (the time period from the first double¬-blind injection of study drug up to the day of last injection + 70 days) were reported.
Groups:
- Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg: Participants, who were receiving atorvastatin 20 mg over-encapsulated tablets orally at baseline, received Alirocumab 75 mg SC injection Q2W, atorvastatin 20 mg over-encapsulated tablets orally QD, and placebo for ezetimibe over-encapsulated tablets orally QD added to stable LMT for 24 weeks. Alirocumab dose up¬-titrated to 150 mg Q2W from Week 12 when LDL-¬C levels ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) at Week 8, based on baseline disease characteristic and medical history.
- Ezetimibe 10 mg + Atorvastatin 40 mg: Participants, who were receiving atorvastatin 40 mg over-encapsulated tablets orally at baseline, received ezetimibe 10 mg over-encapsulated tablets orally QD, atorvastatin 40 mg over-encapsulated tablets orally QD, and placebo for alirocumab SC injection.Q2W added to stable LMT for 24 weeks.
Arm/Group | Atorvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 20 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg | Atorvastatin 80 mg | Rosuvastatin 40 mg | Ezetimibe 10 mg + Atorvastatin 40 mg | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg
Serious Adverse Events (participants affected / at risk) | 2/57 | 5/55 | 3/57 | 4/47 | 2/45 | 2/46 | 1/47
Other Adverse Events (participants affected / at risk) | 17/57 | 24/55 | 15/57 | 18/47 | 23/45 | 12/46 | 19/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin 40 mg (N=57) | Ezetimibe 10 mg + Atorvastatin 20 mg (N=55) | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg (N=57) | Atorvastatin 80 mg (N=47) | Rosuvastatin 40 mg (N=45) | Ezetimibe 10 mg + Atorvastatin 40 mg (N=46) | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg (N=47)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin 40 mg (N=57) | Ezetimibe 10 mg + Atorvastatin 20 mg (N=55) | Alirocumab 75 mg/up to 150 mg + Atorvastatin 20 mg (N=57) | Atorvastatin 80 mg (N=47) | Rosuvastatin 40 mg (N=45) | Ezetimibe 10 mg + Atorvastatin 40 mg (N=46) | Alirocumab 75 mg/up to 150 mg + Atorvastatin 40 mg (N=47)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 3 (6) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 5 (5) | 3 (4) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 5 (6) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (6) | 1 (1) | 4 (4) | 1 (2) | 3 (3) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 2 (3) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 2 (3) | 0 (0) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (6) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 5 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.